CLINICAL TRIAL: NCT00670046
Title: Randomized, Controlled Phase II Study of Valproic Acid in Patients With Non-metastatic Biochemical Progression of Prostate Cancer
Brief Title: Valproic Acid in Treating Patients With Progressive, Non-Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated per the PI decision.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J07122; P30CA068485 (NIH); CDR0000595004; NA_00010227 (Other: JHM IRB)
Record Dates: First submitted 2008-04-30; First posted 2008-05-01 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (standard of care) (Other): Patients undergo observation according to the standard of care. Patients complete quality of life questionnaires at baseline, 6 months, and 1 year.
  Interventions: Other: standard of care follow-up
- Arm II (valproic acid) (Experimental): Patients receive oral valproic acid twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients complete quality of life questionnaires at baseline, 6 months, and 1 year.
  Interventions: Drug: valproic acid

INTERVENTIONS:
Drug: valproic acid — given orally
  Other Names: VPA
  Arms: Arm II (valproic acid)
Other: standard of care follow-up — participant follow the standard of care for patient with metastatic prostate cancer
  Arms: Arm I (standard of care)

SUMMARY:
RATIONALE: Valproic acid may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether valproic acid is more effective than observation in treating patients with prostate cancer.

PURPOSE: This randomized phase II trial is studying how well valproic acid works in treating patients with progressive, non-metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess whether treatment with valproic acid (a type I histone deacetylase inhibitor) can alter the kinetics of prostate-specific antigen (PSA) progression in patients with non-metastatic prostate cancer and biochemical progression.

Secondary

* Determine the duration of PSA response.
* Assess the percentage of patients who achieve a complete response.
* Assess the percentage of patients who achieve a partial response.
* Assess the quality of life of these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 arms.

* Arm I (observation): Patients undergo observation according to standard of care.
* Arm II (valproic acid): Patients receive oral valproic acid twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients complete quality of life questionnaires at baseline, 6 months, and 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * Asymptomatic, non-metastatic disease
* Biochemical progression after definitive local therapy (radical prostatectomy)

  * Most recent prostate-specific antigen (PSA) level ≥ 1.0 ng/mL AND rising over the prior value
  * No clinical or radiological evidence of local progression
* PSA doubling time (DT) < 10 months after local therapy (in patients who have not received prior hormone therapy)

  * At least three PSA values (each at least 4 weeks apart) are required to calculate the PSA-DT
* No clinical or radiological evidence of metastatic disease, including bone metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Total bilirubin normal
* AST/ALT < 2.5 times upper limit of normal
* Creatinine ≤ 2.5 mg/dL
* Platelet count > 125,000/mm^3
* PT and aPTT ≤ 1.3 times above the standard reference
* Albumin ≥ 3.5 g/dL
* Geographically accessible and willing to participate in all stages of study treatment
* No active second malignancy
* No known HIV positivity
* No active, uncontrolled infection (e.g., hepatitis A, B, or C infection)
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to valproic acid
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal study treatment and follow-up
* No history of hepatic disease or significant hepatic dysfunction
* No history of pancreatitis
* No history of seizure disorder or clinically treated bipolar disorder

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior hormone therapy
* No prior valproic acid
* At least 2 weeks since prior drugs specifically known to interact with valproic acid including, but are not limited to, aspirin, felbamate, rifampin, amitriptyline/nortriptyline, carbamazepine, clonazepam, diazepam, ethosuximide, lamotrigine, phenobarbital, primidone, phenytoin, tolbutamide, warfarin, or zidovudine
* No concurrent systemic chemotherapy for prostate cancer
* No other concurrent investigational drugs

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Rodriguez, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Standard of Care) | Arm II (Valproic Acid)
Started | 7 | 8
Completed | 6 | 6
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Standard of Care) | Arm II (Valproic Acid) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Exhibiting an Increase in Observed or Predicted Prostate-specific Antigen (PSA) Doubling Time
Description: Number of participants exhibiting an increase in observed or predicted prostate-specific antigen (PSA) doubling time after initiation of the study. Blood was drawn monthly during study period (1 year), serum PSA was measured & PSADT calculated. A doubling time of > 10 month is defined as complete response (3. Secondary Outcome) and this criteria was based on the Pound et al JAMA 1999, Vol 281(No 17) pgs 1591-1697 paper. Any increase in PSADT is defined as partial response (4. Secondary Outcome).
Time Frame: 1 year
Population: One participant from Arm 1 was lost to follow-up; One participant from Arm II was lost to follow-up and another withdrew consent
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Standard of Care) | Arm II (Valproic Acid)
Number analyzed (Participants) | 6 | 6
Participants | 3 | 5

2. Secondary Outcome: Duration of PSA Response as Assessed by PSA Doubling Time (PSADT)
Description: Serum PSA was measured once a month, each month for the one year the subjects were on the protocol. PSA Doubling time is defined as the duration for PSA levels in the blood to increase by 100 percent, and is calculated based on the rate of change in serum PSA values. Prostate-specific antigen doubling time (PSADT) was calculated by natural log of 2 (0.693) divided by the slope of the relationship between the log of PSA and time of PSA measurement for each patient (Pound et al JAMA 1999, Vol 281(No 17) pgs 1591-1697), therefore it can be much greater than the 12 months that we followed the patients for. PSADT was calculated for pre enrollment, at the mid point of the study & at the end of study.
Time Frame: pre-study, mid-study, end of study (up to 1 year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Arm I (Standard of Care) | Arm II (Valproic Acid)
Number analyzed (Participants) | 6 | 6
months
  Pre-Study | 6.3 (1.9) | 4.0 (2.8)
  Mid-Study | 6.9 (4.0) | 14.1 (9.9)
  End of study | 7.0 (3.8) | 40.7 (46.1)

3. Secondary Outcome: Number of Participants Who Achieve a Complete Response
Description: Complete response was defined as PSA Doubling Time increasing to greater than 10 months. Blood was drawn monthly during study period (1 year), serum PSA was measured & PSADT calculated. The > 10 month criteria was based on the Pound et al JAMA 1999, Vol 281(No 17) pgs 1591-1697 paper.
Time Frame: one year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Standard of Care) | Arm II (Valproic Acid)
Number analyzed (Participants) | 6 | 6
Participants | 1 | 4

4. Secondary Outcome: Number of Participants Who Achieve a Partial Response
Description: Partial Response was defined as any participant that showed an increase in PSA doubling time
Time Frame: one year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Standard of Care) | Arm II (Valproic Acid)
Number analyzed (Participants) | 6 | 6
Participants | 2 | 1

5. Secondary Outcome: Functional Assessment of Cancer Therapy - Prostate (FACT-P) Score
Description: Study questionnaire, known as "Functional Assessment of Cancer Therapy - Prostate (FACT-P), were given to participant to complete during study participation. FACT-P is a validated tool to assess self-perceived functionality, psychosocial well-being, and quality of life; and the scoring of the questionnaire was based on the technique published by FACIT (Functional Assessment of Chronic Illness Therapy). The FACT-P is a 39-item questionnaire, with each item being scored from on a Likert scale of 0-4. The total score ranges from 0-156, with a higher score reflecting a better outcome.
Time Frame: at time of enrollment, mid-study, end of study (up to 1 year)
Population: One participant from Arm 1 was lost to follow-up; One participant from Arm II was lost to follow-up and another withdrew consent; Average FACT-P scores for both arms at Study enrollment, mid study and at end of study is being reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (Valproic Acid)
Number analyzed (Participants) | 6 | 6
units on a scale
  at time of Study Enrollment | 133 (7.5) | 138.5 (5.5)
  Mid Study | 134.8 (4.1) | 126.6 (23.4)
  End of Study | 133.2 (10.3) | 90.4 (42.3)

ADVERSE EVENTS:
Time Frame: One year
Description: AE was self-reported at every study visit and also on-going basis. Participants had access to PI and research nurse at all times during the study.
Arm/Group | Arm I (Standard of Care) | Arm II (Valproic Acid)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

LIMITATIONS AND CAVEATS:
The study was designed to have power with 15 patients in each arm. The study was closed before we reached the target as the PI changed institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes